CLINICAL TRIAL: NCT06466837
Title: Promoting Self-management Behaviours Among Older Adults With Diabetes Mellitus by Integrating Just-In-Time Adaptive Interventions in Mobile Health Applications: A Randomized Controlled Trial
Brief Title: Just-In-Time Adaptive Interventions for Diabetic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Arkers, Wong, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AWong
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Diabetes; Self-Control; Telemedicine
Keywords: telecare; older adults; diabetes
MeSH Terms: conditions — Diabetes Mellitus; Self-Control

STUDY DESIGN:
Intervention Model Description: Single-blinded, two-armed, randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: The research assistant, who will be responsible for data collection, will be masked for the group allocation during the whole process.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Just-in-time Intervention (Experimental): They will receive just-in-time intervention and 3 monthly nursing consultations.
  Interventions: Behavioral: Just-in-time intervention
- Active Control (Active Comparator): They will receive 6 bi-weekly nursing consultations.
  Interventions: Behavioral: Active control

INTERVENTIONS:
Behavioral: Just-in-time intervention — The intervention group participants will receive just-in-time intervention from a developed app for healthy behavior reminder
  Arms: Just-in-time Intervention
Behavioral: Active control — The control group participants will receive six nursing consultations during the 3-month program period.
  Arms: Active Control

SUMMARY:
The addition of proactive nurse consultations was useful to older adults with diabetes mellitus in facilitating their chronic disease self-management. However, the service is time and resource-intensive. With the support of advanced technology, mhealth App seems to be a convenient way to support patients in managing diabetes.

DETAILED DESCRIPTION:
This study examines the effectiveness of mhealth App plus nurse consultations in promoting self-management behaviours for diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* With a confirmed DM diagnosis for one year or more than one year
* Using governmental mhealth App
* Living in an area with Internet coverage

Exclusion Criteria:

* Already engaged in other mHealth programmes
* Physical and cognitive limitations

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | baseline, three-month, and six-month
  Measured using the A1C Now device, with blood drawn from the subjects' finger
Diabetic self-management behaviour | baseline, three-month, and six-month
  measured using the Summary of Diabetes Self-care. Total scores range from 0 to 42, with higher scores representing better self-management performance. Activities questionnaire

SECONDARY OUTCOMES:
Change in quality of life | baseline, three-month, and six-month
  By using the Chinese version of the 12-item Short Form Health Survey. Total score ranges from 0 to 100, higher the better.
  version 2
Change in medication adherence | baseline, three-month, and six-month
  Measure this by using the Adherence to Refills and Medications Scale. Scores from 12 to 48, higher score better medication adherence.
Change in health service utilization | baseline, three-month, and six-month
  Measure the total number of unscheduled visits to general out-patient departments, general practitioners, emergency departments, and hospitals, and the total frequency of health service attendance
Cost | three-month, and six-month
  The cost of the app, including development of new features and maintenance costs, will be estimated from the provider and societal perspectives, including the subjects' travelling costs and time. An ingredient approach will be adopted to estimate the cost.
satisfaction with the JITAIs, as well as usability and technical problems | three-month
  using semi-structured group interviews with the intervention group participants

CONTACTS AND LOCATIONS:
Overall Officials: Arkers Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University; Arkers NR Wong, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- District Health Center, Hong Kong, Hong Kong